CLINICAL TRIAL: NCT04452565
Title: Randomized Controlled Phase 2/3 Clinical Trial of NA-831 Alone or With Atazanavir, or NA-831 With Dexamethasone, or Atazanavir With Dexamethasone in the Treatment of COVID-19 Infection
Brief Title: NA-831, Atazanavir and Dexamethasone Combination Therapy for the Treatment of COVID-19 Infection
Acronym: NATADEX
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biomed Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NATADEX
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Coronavirus Infection; Severe Acute Respiratory Infection; Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: NA-831; Atazanavir; Dexamethasone; COVID-19; Coronavirus Infection; Severe Acute Respiratory Syndrome
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome | interventions — Atazanavir Sulfate; Dexamethasone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active Comparator: NA-831 alone (Active Comparator): Arm 1: NA-831 30 mg orally twice a day for one day, followed by 30 mg once day for four consecutive days (Five days in total). The drug will be supplied in 30 mg capsule
  Interventions: Drug: Drug: NA-831
- Active Comparator: NA-831 plus Atazanavir Sulfate (Active Comparator): Arm 2: NA-831 60 mg orally twice a day for one day, followed by 30 mg once a day for four consecutive days (Five days in total). The drug will be supplied in 30 mg capsule.
  AND Atazanavir 400 mg orally twice a day for one day, followed by 200 mg daily for four consecutive days (five days total). The drug will be supplied in 200 mg tablets.
  Interventions: Combination Product: NA-831 and Atazanavir
- Active Comparator: NA-83 plus Dexamethasone (Active Comparator): Active Comparator: NA-831 30 mg capsule plus Dexamethasone 4 mg Arm 3: NA-831 60 mg orally twice a day for one day, followed by 30 mg once a day for four consecutive days (Five days in total). The drug will be supplied in 30 mg capsule.
  AND Dexamethasone 8 mg orally twice a day for one day, followed by 4 mg daily for four consecutive days (five days total). The drug will be supplied in 4 mg tablets.
  Interventions: Combination Product: NA-831and Dexamethasone
- Active Comparator: Atazanavir and Dexamethasone (Active Comparator): Atazanavir 400 mg orally twice a day for one day, followed by 200 mg daily for four consecutive days (five days total). The drug will be supplied in 200 mg tablets.
  AND Dexamethasone 8 mg orally twice a day for one day, followed by 4 mg daily for four consecutive days (five days total). The drug will be supplied in 4 mg tablets.
  Interventions: Combination Product: Atazanavir and Dexamethasone

INTERVENTIONS:
Drug: Drug: NA-831 — NA-831 is a neuroprotective drug, available at 30 mg capsule
  Arms: Active Comparator: NA-831 alone
Combination Product: NA-831 and Atazanavir — Drug: NA-831 Neuroprotective drug Other Name: Traneurocin 30 mg capsule
  Drug: Atazanavir Sulfate Antiviral drug Other Name: Atazanavir Sulfate 200 mg tablet
  Other Names: and Atazanavir
  Arms: Active Comparator: NA-831 plus Atazanavir Sulfate
Combination Product: NA-831and Dexamethasone — Drug: NA-831 Neuroprotective drug Other Name: Traneurocin 30 mg capsule
  Drug: Dexamethasone anti-inflammatory drug Other Name: Dexamethasone 4 mg
  Other Names: Dexamethasone
  Arms: Active Comparator: NA-83 plus Dexamethasone
Combination Product: Atazanavir and Dexamethasone — Drug: Atazanavir Sulfate Antiviral drug Other Name: Atazanavir Sulfate 200 mg tablet Drug: Dexamethasone anti-inflammatory drug Other Name: Dexamethasone 4 mg
  Other Names: Dexamethasone
  Arms: Active Comparator: Atazanavir and Dexamethasone

SUMMARY:
This Phase 2/3 trial evaluates four treatment strategies for non-critically ill hospitalized participants (not requiring ICU admission and/or mechanical ventilation) with SARS CoV-2 infection, in which participants will receive NA-831 or Atazanavir with or without Dexamethasone.

DETAILED DESCRIPTION:
The clinical Phase 2/3 evaluates the safety and efficacy of NA-831 alone, and a combination therapy comprises NA-831 with an anti-viral drug Atazanavir, NA-831 with an anti-inflammatory drug, Dexamethasone and a potential synergy between Atazanavir and Dexamethasone. NA-831 is also known as Traneurocin is a neuroprotective drug that is in clinical study for the treatment of Alzheimer's Disease. Participants will receive NA-831 or Atazanavir with or without Dexamethasone. Investigators are primarily interested in the time to recovery. In addition to study medications there will be daily symptom surveys for 14 days, then weekly thereafter for 3 weeks resulting in a total duration of follow up of 36 days. During hospitalization, daily symptom surveys will be carried out in conjunction with the study coordinators. Upon discharge participants will have the option to complete electronic symptom surveys or complete symptom surveys via telephone with the study coordinator. If electronic symptom surveys are selected on discharge participants will also receive a follow-up call from a study coordination every 7 days during the initial 14 day period. In addition, failure to submit a symptom survey will prompt a study follow up call.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for management of SARS CoV-2 infection
* Positive SARS CoV-2 test
* Age > = 18 years
* Provision of informed consent
* Electrocardiogram (ECG) ≤ 48 hours prior to enrollment
* Complete blood count, glucose-6 phosphate-dehydrogenase (G6PD), comprehensive metabolic panel and magnesium ≤ 48 hours prior to enrollment from standard of care.
* If participating in sexual activity that could lead to pregnancy, individuals of reproductive potential who can become pregnant must agree to use contraception throughout the study. At least one of the following must be used throughout the study:

  * Condom (male or female) with or without spermicide
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Hormone-based contraceptive

Exclusion Criteria:

* Contraindication or allergy to NA-831, Atazanavir, Dexamethasone
* Current use any antiviral drug or anti-inflammatory drug
* Concurrent use of another investigational agent
* Invasive mechanical ventilation
* Participants who have any severe and/or uncontrolled medical conditions such as:

  * unstable angina pectoris,
  * symptomatic congestive heart failure,
  * myocardial infarction,
  * cardiac arrhythmias or know prolonged QTc > 470 males, > 480 female on ECG
  * pulmonary insufficiency,
  * epilepsy (interaction with chloroquine),
* Prior retinal eye disease
* Concurrent malignancy requiring chemotherapy
* Known Chronic Kidney disease, eGFR < 10 or dialysis
* G-6-PD deficiency, if unknown requires G6PD testing prior to enrollment

  * Known Porphyria
  * Known myasthenia gravis
  * Currently pregnant or planning on getting pregnant while on study
  * Breast feeding
  * AST/ALT > five times the upper limit of normal ULN
  * Bilirubin > five times the ULN
  * Magnesium < 1.4 mEq/L
  * Calcium < 8.4 mg/dL > 10.6 mg/dL
  * Potassium < 3.3 > 5.5 mEg/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
1. Time (Hours) to recovery | [ Time Frame: 36 days ]
  Time (hours) from randomization to recovery defined as 1) absence of fever, as defined as at least 48 hours since last temperature ≥ 38.0°C without the use of fever-reducing medications AND 2) absence of symptoms of greater than mild severity for 24 hours AND 3) not requiring supplemental oxygen beyond pre-COVID baseline AND 4) freedom from mechanical ventilation or death

SECONDARY OUTCOMES:
Time fever resolution | [ Time Frame: 36 days ]
  Time to resolution of fever defined as at least 48 hours since last temperature ≥ 38.0°C without the use of fever-reducing medications

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Tran, PhD, Study Director — Biomed Industries, Inc.
Locations (30):
- United States (30):
  - Coronavirus Research Institute- Testing Site, Los Angeles, California
  - Coronavirus Research Institute, Orange, California
  - Coronavirus Research Institute-Testing Site, Palo Alto, California
  - Coronavirus Research Institute-Testing Site, Sacramento, California
  - Coronavirus Research Institute-Testing Site, San Diego, California
  - Coronavirus Research Testing Site, San Francisco, California
  - Coronavirus Research Institute-Testing Site, Sunnyvale, California
  - Coronavirus Research Institute-Testing Site, Washington D.C., District of Columbia
  - Coronavirus Research Institute-Testing Site, Fort Lauderdale, Florida
  - Coronavirus Research Institute-Testing Site, Tampa, Florida
  - Coronavirus Research Institute- Testing Site, Chicago, Illinois
  - Coronavirus Research Institute-Testing Site, Naperville, Illinois
  - Coronavirus Research Institute-Testing Site, Baltimore, Maryland
  - Coronavirus Research Institute-Testing Site, Bethesda, Maryland
  - Coronavirus Research Institute-Testing Site, Boston, Massachusetts
  - Coronavirus Research Institute-Testing Site, Worcester, Massachusetts
  - Coronavirus Research Institute-Testing Site, Ann Arbor, Michigan
  - Coronavirus Research Institute-Testing Site, Detroit, Michigan
  - Coronavirus Research Institute-Testing Site, Newark, New Jersey
  - Coronavirus Research Institute-Testing Site, New York, New York
  - Coronavirus Research Institute- Testing Site, Rochester, New York
  - Coronavirus Research Institute-Testing Site-, The Bronx, New York
  - Coronavirus Research Institute-Testing Site, Durham, North Carolina
  - Coronavirus Research Institute-Testing Site, Philadelphia, Pennsylvania
  - Coronavirus Research Institute- Testing Site, Fort Sam Houston, Texas
  - Coronavirus Research Institute-Testing Site, Galveston, Texas
  - Coronavirus Research Institute-Testing Site, Houston, Texas
  - Coronavirus Research Institute-Testing Site, Kirkland, Washington
  - Coronavirus Research Institute-Testing Site, Seattle, Washington
  - Coronavirus Research Institute-Testing Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No